CLINICAL TRIAL: NCT03849443
Title: Single Versus Multi-Dose Oral and Intravenous Tranexamic Acid in Patients at High Risk for Blood Transfusion After Spine Surgery
Brief Title: Single Versus Multi-Dose Oral and Intravenous Tranexamic Acid Patients at High Risk for Blood Transfusion After Spine Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17081704-IRB01; NCT04672213 (obsolete NCT alias)
Record Dates: First submitted 2018-11-30; First posted 2019-02-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Open Posterior Thoracolumbar Spinal Fusion Procedure
MeSH Terms: interventions — Ascorbic Acid; Tablets; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1 PLACEBO (Placebo Comparator)
  Interventions: Drug: Vitamin C 250 MG Oral Tablet
- Group 2 IV TXA (Experimental)
  Interventions: Drug: Tranexamic Acid Injectable Product (1000 mg intravenous bolus); Drug: Vitamin C 250 MG Oral Tablet
- Group 3 Pre-Oral TXA (Experimental)
  Interventions: Drug: Vitamin C 250 MG Oral Tablet; Drug: Tranexamic Acid 650Mg Tablet
- Group 4 Full Oral TXA (Experimental)
  Interventions: Drug: Tranexamic Acid 650Mg Tablet

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Product (1000 mg intravenous bolus) — Intravenous methods to decrease blood loss
  Arms: Group 2 IV TXA
Drug: Vitamin C 250 MG Oral Tablet — Oral method of placebo
  Arms: Group 1 PLACEBO; Group 2 IV TXA; Group 3 Pre-Oral TXA
Drug: Tranexamic Acid 650Mg Tablet — Oral method of treatment group
  Arms: Group 3 Pre-Oral TXA; Group 4 Full Oral TXA

SUMMARY:
As tranexamic acid (TXA) becomes more prevalent, all patients are receiving the same dose and method of delivery regardless of their pre-operative risk of transfusion. Therefore, the aim of the study is to determine whether or not repeated dosing of oral or different method of delivery like intravenous (IV) TXA reduces the postoperative reduction in hemoglobin, hematocrit, number of transfusions, and postoperative blood loss following open spine surgery. The regimen that utilizes multiple doses of oral TXA will significantly minimize post-operative blood loss and transfusion requirements compared to the use of a single dose regimen. Furthermore, oral TXA will be as efficacious as intravenous delivery of TXA.

DETAILED DESCRIPTION:
Background/Scientific review:

Open lumbar spine surgery is associated with the risk of moderate to significant blood loss. Because TXA has been shown to significantly reduce the need for blood products during total joint replacement, it is now the standard of care for these procedures at many institutions.1-3 Oral and IV TXA have been found to be similarly efficacious in total joint replacements, but oral TXA is cheaper and allows for ease of repeat dosing.1 Although low preoperative hemoglobin is a risk factor for transfusion, no studies that have compared standard single-dose oral or IV TXA dosing to repeated oral dosing of TXA in patients undergoing open spine surgery.

Study Design: Prospective, randomized, double-blinded study Inclusion Criteria: Any patient older than 18 years old and scheduled for an open posterior thoracolumbar spinal fusion procedure

Exclusion Criteria: Allergy to TXA, acquired disturbances of color vision, refusal of blood products, pre-op use of anticoagulant therapy within five days before surgery, a history of arterial or venous thromboembolic disease (such as DVT, PE, CVA, TIA), pregnancy, breastfeeding, major comorbidities (such as severe ischemic heart disease [New York Heart Association Class III or IV], previous myocardial infarction, severe pulmonary disease, renal impairment, or hepatic failure), patients who decline to participate, intolerance or sensitivity to Vitamin C.

Screening Procedures and Randomization: At the pre-operative clinic appointment and before the day of surgery, the study staff will assess the potential subject's eligibility, which would include asking for any intolerance/sensitivity to Vitamin C. Once eligibility is established, the potential subject will be approached regarding their participation in this clinical trial. The investigators will provide 48 hours before the date of surgery to allot for questions and consideration of the Informed Consent document. Once all patient questions have been answered patients willing to be in the study will sign the Informed Consent. Patients will be randomized, via standard randomization tables that provide a 1:1:1:1 distribution of subjects between the four groups through blocked randomization, no later than the morning of surgery to either of the four treatment groups: Placebo, Preoperative IV TXA, Preoperative-oral TXA only, or Full (pre-op and post-op) Oral TXA.

Sample Size Calculation: Sample size calculation determined that 151 patients per treatment group (604 patients total) are required to provide an alpha of 0.05 and beta of 0.80. This total of 604 patients includes a 10% drop-out rate to allow for protocol deviations.

Demographics/Patient Specifics: Age, sex, ASA score, weight, height, estimated intra-operative blood loss, intra-operative fluids (crystalloid, colloid), operative time, hospitalization days, BMI, pre-operative hemoglobin, hematocrit, PT/INR, PTT, and platelet count.

Treatment Groups:

Group 1 PLACEBO: three 250 mg tablets of ascorbic acid 2 hours prior to incision, placebo IV at time of incision intraoperatively, three 250 mg tablets of ascorbic acid given each day for three days postoperatively (while in the hospital as an inpatient).

Group 2 IV TXA: three 250 mg tablets of ascorbic acid 2 hours prior to incision, 1g IV TXA bolus at time of incision intraoperatively, three 250 mg tablets of ascorbic acid given each day for three days postoperatively (while in the hospital as an inpatient).

Group 3 Pre-Oral TXA: three 625mg tablets of oral TXA 2 hours prior to incision, placebo IV at time of incision intraoperatively, and three 250 mg tablets of ascorbic acid given each day for three days postoperatively (while in the hospital as an inpatient).

Group 4 Full Oral TXA: three 625mg tablets of oral TXA 2 hours prior to incision, placebo IV at time of incision intraoperatively, three 625mg tablets of oral TXA given each day for three days postoperatively (while in the hospital as an inpatient).

Outcome Measurements: (Assessed during hospital stay and at routine outpatient follow-up visit which occurs about 3 weeks after discharge and within 30 days of surgery) Number of patients transfused (primary outcome) and units transfused Post-operative reduction in hemoglobin and hematocrit

Postoperative blood loss will be determined primarily by the postoperative drop in hemoglobin, which is calculated as the patient's preoperative hemoglobin minus the patient's lowest postoperative hemoglobin. Secondarily, postoperative blood and hemoglobin loss will be calculated as a function of patient characteristics including sex, weight, and height as well as preoperative and postoperative hemoglobin balance, using the formulas previously described by Nadler et al and Good et al,5,6 which have been used in prior TXA studies.1,4 Cost comparison - Cost differences resulted from differences in the blood transfusion rate, length of hospital stay, and management of complications as well as from the cost of the TXA itself Complications - DVT/PE, return to the OR within 30 days, superficial or deep infection, and cerebrovascular accident, transient ischemic attack or MI

ELIGIBILITY:
Inclusion Criteria:

* Any patient older than 18 years old
* Scheduled for an open posterior thoracolumbar spinal fusion procedure

Exclusion Criteria:

* Allergy to TXA
* Acquired disturbances of color vision
* Refusal of blood products
* Pre-op use of anticoagulant therapy within five days before surgery
* History of arterial or venous thromboembolic disease (such as DVT, PE, CVA, TIA)
* Pregnancy
* Breastfeeding
* Severe ischemic heart disease [New York Heart Association Class III or IV]
* Previous myocardial infarction
* Severe pulmonary disease
* Renal impairment
* Hepatic failure
* Patients who decline to participate
* Intolerance or sensitivity to Vitamin C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative blood loss | During hospital stay and at routine outpatient follow-up visit which occurs about 3 weeks after discharge and within 30 days of surgery

SECONDARY OUTCOMES:
preoperative and postoperative hemoglobin balance | During hospital stay and at routine outpatient follow-up visit which occurs about 3 weeks after discharge and within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bryce Basques, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data (IPD)

REFERENCES:
- [Result] Fillingham YA, Kayupov E, Plummer DR, Moric M, Gerlinger TL, Della Valle CJ. The James A. Rand Young Investigator's Award: A Randomized Controlled Trial of Oral and Intravenous Tranexamic Acid in Total Knee Arthroplasty: The Same Efficacy at Lower Cost? J Arthroplasty. 2016 Sep;31(9 Suppl):26-30. doi: 10.1016/j.arth.2016.02.081. Epub 2016 Mar 19. PMID 27113948
- [Result] Irwin A, Khan SK, Jameson SS, Tate RC, Copeland C, Reed MR. Oral versus intravenous tranexamic acid in enhanced-recovery primary total hip and knee replacement: results of 3000 procedures. Bone Joint J. 2013 Nov;95-B(11):1556-61. doi: 10.1302/0301-620X.95B11.31055. PMID 24151279
- [Result] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Result] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Result] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Result] Good L, Peterson E, Lisander B. Tranexamic acid decreases external blood loss but not hidden blood loss in total knee replacement. Br J Anaesth. 2003 May;90(5):596-9. doi: 10.1093/bja/aeg111. PMID 12697586